CLINICAL TRIAL: NCT03204071
Title: COMPARATIVE EVALUATION OF SUBGINGIVALLY DELIVERED 1% METFORMIN AND ALOE VERA GEL IN TREATMENT OF INTRABODY DEFECTS IN CHRONIC PERIODONTITIS SUBJECTS: A RANDOMIZED CONTROLLED CLINICAL TRIAL
Brief Title: Locally Delivered Metformin and Aloe Vera for Treatment of Intrabody Defects in Chronic Periodontitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, professor, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/2/2015-2016IG
Record Dates: First submitted 2017-06-28; First posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Group 1 (Placebo Comparator): Placebo gel without active ingredient to be delivered at baseline, 6 and 12 months.
  Interventions: Drug: placebo gel
- Group 2 (Active Comparator): Aloe vera gel to be delivered at baseline, 6 and 12 months.
  Interventions: Drug: Aloevera
- Group 3 (Active Comparator): 1% metformin gel to be delivered at baseline, 6 and 12 months.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: placebo gel — Oral prophylaxis followed by Placebo gel to be delivered in intrabody sites of chronic periodontitis subjects.
  Other Names: inactive drug
  Arms: Group 1
Drug: Aloevera — Oral prophylaxis followed by placement of aloevera gel
  Other Names: AV
  Arms: Group 2
Drug: Metformin — Oral prophylaxis followed by placement of metformin gel
  Other Names: MF
  Arms: Group 3

SUMMARY:
Metformin (MF), a biguanide group of anti-diabetic drug has been shown to enhance osteoblasts differentiation and inhibit osteoclast differentiation in vitro, thus may exhibit a favorable effect on alveolar bone.

AloeVera Gel had also been used in dentistry and showed good results.The present study aims to explore the efficacy of 1% MF gel and aloe vera gel as a local drug delivery system in adjunct to scaling and root planing (SRP) for the treatment of subjects with chronic periodontitis (CP) with intrabody defects.

DETAILED DESCRIPTION:
Aim: To compare the efficacy of locally delivered 1% MF gel and aloe vera gel in treatment of intrabony defects in chronic periodontitis subjects and compare it with placebo gel.

Methods: Ninety subjects were categorized into three treatment groups: Placebo, aloevera gel(AV) and 1% Metformin (MF)after Scaling and root planning (SRP). Clinical parameters were recorded at baseline, 6 and 12 months; they included plaque index (PI), modified sulcus bleeding index (mSBI), pocket probing depth (PPD), and clinical attachment level (CAL). Radiologic assessment of intra-bony defect (IBD) and percentage defect depth reduction (DDR%) was done at baseline, 6 months and 12 months interval using computer-aided software Results: Mean PPD reduction and mean CAL gain was found to greater in MF group than AV and placebo group at all visits. The DDR% was greater in MF group as compared to AV and placebo group.

Conclusion: There was a greater decrease in mSBI and PPD and more CAL gain at the sites treated with AV and MF as an adjunct to SRP in chronic periodontitis subjects with intrabony defects as compared to placebo. The significant IBD depth reduction effect was seen in case of MFgroup.

ELIGIBILITY:
Inclusion Criteria:

Systemically healthy patients with sites showing PPD ≥ 5 mm, CAL ≥ 4 mm and vertical bone loss ≥ 3 mm on intraoral periapical radiographs, with no history of periodontal therapy in the last 6 months.

-

Exclusion Criteria:

* Subjects allergic to MF or AV Those on systemic MF or AV therapy Subjects with aggressive periodontitis Immunocompromised subjects Use of tobacco in any form, alcoholics Lactating, and pregnant females

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change in Bone defect fill | baseline - 6 months & baseline -12 months
  Assessed in percentage

SECONDARY OUTCOMES:
Change in modified sulcus bleeding index | baseline, 6 & 12 months
  scale 0-3
Change in Plaque index | baseline, 6 & 12 months
  scale 0-3
Change in pocket probing depth | baseline, 6 & 12 months
  measured in mm
Clinical attachment level | baseline, 6 & 12 months
  measured in mm